CLINICAL TRIAL: NCT03133468
Title: A First-in-Human, Randomised, Double Blind, Placebo Controlled, Single and Multiple Ascending Oral Dose Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AJM347 in Healthy Male Caucasian and Japanese Subjects in the Fasted and Fed State
Brief Title: Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of AJM347 in Healthy Male Caucasian and Japanese Subjects in the Fasted and Fed State
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EA Pharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: AJM347/CP1; 2017-000259-17 (EudraCT Number); 1009306/8349634 (Other: Covance Clinical Research Unit)
Record Dates: First submitted 2017-04-25; First posted 2017-04-28 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-07

CONDITIONS: Healthy Participants
Keywords: AJM347; pharmacokinetics; food effect study; pharmacodynamics

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Part 1: AJM347 (Experimental): Caucasian and Japanese participants will be randomized to receive one of eight and four single oral doses of AJM347, respectively, administered in the fasted state on Day 1.
  Interventions: Drug: AJM347
- Part 1: Placebo (Placebo Comparator): Caucasian and Japanese participants will be randomized to receive one of eight and four single oral doses of matching placebo, respectively, administered in the fasted state on Day 1.
  Interventions: Drug: Placebo
- Part 2: Low-dose AJM347 (Experimental): Caucasian and Japanese participants will receive a "low" dose of AJM347 (at different frequencies and in either a fed or fasted state) on Day 1 of each of 6 sequential treatment periods.
  Interventions: Drug: AJM347
- Part 2: High-dose AJM347 (Experimental): Caucasian and Japanese participants will receive a "high" dose of AJM347 (at different frequencies and in either a fed or fasted state) on Day 1 of each of 2 sequential treatment periods (the frequency and timing with respect to meals will be determined after review of the data from the low-dose AJM347 groups).
  Interventions: Drug: AJM347
- Part 3: AJM347 (Experimental): Caucasian and Japanese participants will be randomized to receive one of three single doses of AJM347 on the morning of Day 1 and multiple daily doses beginning on the morning of Day 3, with the last dose received on the evening of Day 9. The actual doses, dosing frequencies, and timings with respect to meals to be employed in Part 3 of the study will be determined after review of the data from dose groups in Parts 1 and 2 of the study.
  Interventions: Drug: AJM347
- Part 3: Placebo (Placebo Comparator): Caucasian and Japanese participants will be randomized to receive one of three single doses of matching placebo on the morning of Day 1 and multiple daily doses beginning on the morning of Day 3, with the last dose received on the evening of Day 9. The actual doses, dosing frequencies, and timings with respect to meals to be employed in Part 3 of the study will be determined after review of the data from dose groups in Parts 1 and 2 of the study.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AJM347 — Oral administration
  Arms: Part 1: AJM347; Part 2: High-dose AJM347; Part 2: Low-dose AJM347; Part 3: AJM347
Drug: Placebo — Oral administration
  Arms: Part 1: Placebo; Part 3: Placebo

SUMMARY:
This study will be conducted to determine the safety and tolerability of single and multiple oral ascending doses of AJM347 in healthy male participants, and to assess the pharmacodynamic response following single and multiple oral ascending doses of AJM347 in the same population. This study will also aim to determine the single and multiple oral ascending dose pharmacokinetics of AJM347 and its metabolite in healthy male participants, and to determine the effect of food on the single and multiple oral dose pharmacokinetics of AJM347 and its metabolite in the same population.

ELIGIBILITY:
Inclusion Criteria:

Main Inclusion Criteria for all participants:

* Participants will be male
* Participants will be in good health

Main Inclusion Criteria for Japanese participants:

* Be ≥20 to ≤45 years of age
* Have body mass index (BMI) ≥18.5 to ≤25.0 kilograms per meters squared (kg/m^2)
* Be Japanese

Main Inclusion Criteria for Caucasian participants:

* Be ≥18 to ≤45 years of age
* Have a BMI ≥18.5 to ≤30.0 kg/m^2
* Be Caucasian

Exclusion Criteria:

Main Exclusion Criteria for all participants:

Participants will be excluded from the study if they satisfy any of the following criteria at the Screening visit, unless otherwise stated.

* Participants who have donated or lost ≥200 milliliters (mL) blood within 1 month or ≥400 mL within 3 months prior to Check-in
* Participants who have an abnormality in heart rate, blood pressure, temperature, or respiration rate at Screening
* Participants who have:

  * a positive urine drugs of abuse screen;
  * a positive alcohol breath test
* Participants who have an abnormality in the 12-lead electrocardiogram (ECG) at Screening
* Participants who are still participating in another clinical study (eg, attending follow-up visits) or who have participated in a clinical study involving administration of an investigational drug (new chemical entity) in the past 3 months prior to first dose administration
* Participants who have a significant history of drug allergy, as determined by the Investigator
* Participants who have any clinically significant abnormal physical examination finding
* Participants who:

  * are carriers of the hepatitis B surface antigen (HBsAg);
  * are carriers of the hepatitis C antibody;
  * have a positive result for the test for human immunodeficiency virus (HIV) antibodies
* Participants who, in the opinion of the Investigator, should not participate in this study

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2017-07-25 (Actual); Primary Completion 2018-07-06 (Actual); Study Completion 2018-07-06 (Actual)

PRIMARY OUTCOMES:
Number of participants with any adverse event (AE) | Part 1, up to Days 7 to 9; Part 2, up to Days 7 to 9; Part 3, up to Day 15 (Parts 1, 2, and 3 are not continuous)
  An AE is any untoward medical occurrence in a patient or clinical investigation participant administered an investigational product. An AE does not necessarily have a causal relationship with the medicinal product.

SECONDARY OUTCOMES:
Number of participants with abnormal, clinically significant physical examination findings | Part 1, up to Days 7 to 9; Part 2, up to Days 7 to 9; Part 3, up to Day 15 (Parts 1, 2, and 3 are not continuous)
  Clinical significance will be determined by the investigator.
Number of participants with abnormal, clinically significant vital sign values | Part 1, up to Days 7 to 9; Part 2, up to Days 7 to 9; Part 3, up to Day 15 (Parts 1, 2, and 3 are not continuous)
  Clinical significance will be determined by the investigator.
Number of participants with abnormal, clinically significant 12-lead electrocardiogram (ECG) values | Part 1, up to Days 7 to 9; Part 2, up to Days 7 to 9; Part 3, up to Day 15 (Parts 1, 2, and 3 are not continuous)
  Clinical significance will be determined by the investigator.
Number of participants with abnormal, clinically significant clinical laboratory values | Part 1, up to Days 7 to 9; Part 2, up to Days 7 to 9; Part 3, up to Day 15 (Parts 1, 2, and 3 are not continuous)
  Clinical significance will be determined by the investigator.
Mean plasma concentrations of AJM347 and its metabolite | Part 1, Days 1 to 3; Part 2, Days 1 to 3; Part 3, Days 1 to 3, Day 7, Days 9 to 11 (Parts 1, 2, and 3 are not continuous)
  Blood samples will be collected at the specified time points for the determination of plasma concentrations of AJM347 and its metabolite.
Mean urinary concentrations of AJM347 and its metabolite | Part 1, Days 1 to 3; Part 3, Days 1 to 10
  Urine samples will be collected at the specified time points for the determination of urine concentrations of AJM347 and its metabolite.
Inhibition rate of ligand-binding activity | Part 1, Days 1 and 2; Part 3, Days 1 and 2, Days 7, 9, and 10
  The rate of inhibition of ligand-protein binding will be measured.

CONTACTS AND LOCATIONS:
Locations (1):
- Covance Clinical Research Unit (CRU) Ltd, Leeds, United Kingdom

IPD SHARING:
Plan to Share IPD: No